CLINICAL TRIAL: NCT05037149
Title: Ph.1, Open-Label, Dose Escalation & Expansion for Safety, Tolerability, PK, & Anti-Tumor Activity of STP707 Administered IV in Subjects With Advanced/Metastatic or Surgically Unresectable Solid Tumors Who Are Refractory to Standard Therapy.
Brief Title: Ph. 1, Evaluation of Safety, Tolerability, PK, Anti-tumor Activity of STP707 IV in Subjects With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-707-001
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: One subject will be enrolled at dose level 1. After the first subject has passed the DLT period, defined as 28 days, the second and third subject will be enrolled at least 24 hours apart. If more than 3 subjects have been identified for a given dose level, additional subjects may be enrolled in a lower dose level that has passed the DLT period up to a maximum of 12 subjects per dose level for dose levels 3 and 4 and up to a maximum of 9 subjects for dose levels A and 5. Subjects enrolled to backfill cohorts may be enrolled simultaneously, without a waiting period between subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1: Arm A (Experimental): Cohort 1: STP707 3 mg dose IV infusion, administered on D1,D8,D15,D22 of a 28-Day cycle. If the patient is deriving clinical benefit from the agent it maybe continued and administered on D1,D8, D15 and D22 for each successive cycle.
  Interventions: Drug: STP707
- Part 1: Arm B (Experimental): Cohort 2: STP707 6 mg dose IV infusion, administered on D1,D8,D15,D22 of a 28-Day cycle. If the patient is deriving clinical benefit from the agent it maybe continued and administered on D1,D8, D15 and D22 for each successive cycle.
  Interventions: Drug: STP707
- Part 1: Arm C (Experimental): Cohort 3: STP707 12 mg dose IV infusion, administered on D1,D8,D15,D22 of a 28-Day cycle. If the patient is deriving clinical benefit from the agent it maybe continued and administered on D1,D8, D15 and D22 for each successive cycle.
  Interventions: Drug: STP707
- Part 1: Arm D (Experimental): Cohort 4: STP707 24 mg dose IV infusion, administered on D1,D8,D15,D22 of a 28-Day cycle. If the patient is deriving clinical benefit from the agent it maybe continued and administered on D1,D8, D15 and D22 for each successive cycle.
  Interventions: Drug: STP707
- Part 1: Arm E (Experimental): Cohort A: STP707 36 mg dose IV infusion, administered on D1,D8,D15,D22 of a 28-Day cycle. If the patient is deriving clinical benefit from the agent it maybe continued and administered on D1,D8, D15 and D22 for each successive cycle.
  Interventions: Drug: STP707
- Part 1: Arm F (Experimental): Cohort 5: STP707 48 mg dose IV infusion, administered on D1,D8,D15,D22 of a 28-Day cycle. If the patient is deriving clinical benefit from the agent it maybe continued and administered on D1,D8, D15 and D22 for each successive cycle.
  Interventions: Drug: STP707

INTERVENTIONS:
Drug: STP707 — STP707 Powder for Injection
  Other Names: STP707 Powder for Injection

SUMMARY:
An open label, dose escalation and dose expansion study to evaluate the safety, tolerability, and anti-tumor activity of STP707 with IV administration in subjects with advanced/metastatic or surgically unresectable solid tumors who are refractory to standard therapy.

DETAILED DESCRIPTION:
A phase 1, open label, dose escalation and dose expansion study to evaluate the safety, tolerability, and anti-tumor activity of STP707 with IV administration in subjects with advanced/metastatic or surgically unresectable solid tumors who are refractory to standard therapy.

The primary objective of this study is to determine the MTD or RP2D of STP707 and to establish the dose of STP707 recommended for future phase 2 studies administered intravenously.

A total of 30 subjects will be enrolled in dose escalation. Once MTD or RP2D has been established, up to 10 additional subjects will enrolled to confirm safety and explore anti-tumor activity.

Up to 5 dose levels will be explored (3,6,12,24,48 mg dose levels). Intermediate doses between scheduled dose levels maybe explored during escalation. A cycle is 28 days.

Dose escalation will follow a standard 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed advanced / metastatic or surgically unresectable solid tumors whose tumors are refractory to standard therapy
2. Measurable disease per RECIST v 1.1 (primary or metastatic disease)
3. ECOG performance status 0 - 1
4. Life expectancy of at least 3 months
5. Age ≥18 years
6. Signed, written Institutional Review Board (IRB) approved informed consent
7. A negative serum pregnancy test (for nonsterile women of child-bearing potential)
8. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal
   * AST (SGOT), ALT (SGPT) ≤ 5 times upper limit of normal because of cancer or metastases to the liver
9. Acceptable renal function, defined as:

   o Serum creatinine ≤ 1.5 ULN or Creatinine Clearance ≥ 50 mL/minute
10. Acceptable hematologic status:

    * Hemoglobin ≥ 9 g/dL (a transfusion is allowed if Hemoglobin stays stable thereafter)
    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
    * Platelet count ≥ 100,000 plt/mm3 x 109/ L
11. Urinalysis with no clinically significant abnormalities
12. Acceptable coagulation status with partial thromboplastin time (PTT) and International Normalized Ratio (INR) ≤ 1.5 times upper limit of normal unless patient is on anticoagulants and has stable PTT and PT that are within normal therapeutic range for disease under management
13. Subject has adequate vitamin D level, as defined by serum total 25-Hydroxyvitamin D [25(OH)D] ≥ 20 to < 60 ng/mL. If subjects are below this threshold, they may receive vitamin D supplementation se per clinic dosing guidelines and may still be enrolled provided they are started on vitamin D supplementation
14. Completion of all previous treatments (including surgery, systemic chemotherapy, and radiotherapy) at least 3 weeks before screening
15. For men and women of child-producing potential, the use of effective contraceptive methods during the study

Exclusion Criteria:

1. Baseline Q-T corrected interval (QTc) interval of > 470 msec for all subjects calculated using Fridericia's formula
2. New York Heart Association Class III or IV cardiac disease, or myocardial infarction, severe unstable angina, coronary/peripheral artery bypass graft, congestive heart failure within the past 6 months
3. Known active, uncontrolled infection with HIV or hepatitis B; subjects with hepatitis B allowed if on anti-viral therapy and have a viral load ≤ 500 IU; patients with a history of HIV must be on antiretroviral therapy for at least four weeks and have an HIV viral load ≤ 400 copies/mL, have CD4+ T cell counts ≥ 350 cells/uL and no history of AIDS-defining opportunistic infections within 3 months prior to treatment
4. Major surgical procedure within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure, during the course of the study. (Note: Placement of a central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure.)
5. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
6. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Participation in a clinical study involving administration of an investigational compound within the past 30 days prior to study entry.
8. Unwillingness or inability to comply with procedures required in this protocol
9. Known allergy or hypersensitivity to the study drug(s) or one of the ingredients in the formulation (e.g., Trehalose dihydrate)
10. Existence of any surgical, medical or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Day Cycle
  Recommended starting dose & schedule
Limited Dose Toxicity (LDT) | 28 day cycle
  Recommended starting dose & dose escalation

CONTACTS AND LOCATIONS:
Overall Officials: Andrae Vandross, MD, Principal Investigator — NEXT Oncology; Jason Henry, MD, Principal Investigator — Sarah Cannon Research Institute at HealthONE; Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California; Angela Alistar, MD, Principal Investigator — Atlantic Health System; Hani Babiker, MD, Principal Investigator — Mayo Clinic; Michael Cecchini, MD, Principal Investigator — Yale University; Conor Steuer, MD, Principal Investigator — Emory University; Christina Wu, MD, Principal Investigator — Mayo Clinic; Zhaohui Jin, MD, Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - Mayo Clinic, Phoenix, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - NEXT Oncology, Austin, Texas